CLINICAL TRIAL: NCT02026661
Title: Effectiveness of Intracytoplasmic Sperm Injection and Laser Assisted Hatching on in Vitro Fertilization Outcomes of Patients With Different Causes of Infertility
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 102160-E
Record Dates: First submitted 2014-01-01; First posted 2014-01-03 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- those that did not receive ICSI or LAH
- those that received ICSI only
- those that received LAH only
- those that received both ICSI and LAH

SUMMARY:
To determine the association of factors affecting the clinical pregnancy and live birth rates in patients undergoing in vitro fertilization (IVF) who received intracytoplasmic sperm injection (ICSI) and/or laser assisted hatching (LAH) or neither.

After applying the inclusion and exclusion criteria, a total of 400 women who underwent IVF between January 2007 and December 2010 were included in the analysis. Patients were divided into 4 groups; 1) those that did not receive ICSI or LAH, 2) those that received ICSI only, 3) those that received LAH only, and 4) those that received both ICSI and LAH. Univariate and multivariate analyses were performed.

ELIGIBILITY:
Inclusion Criteria:

* The present study was a retrospective review of the outcomes of women who underwent IVF with or without intracytoplasmic sperm injection (ICSI) at the Far Eastern Memorial Hospital, Taipei, Taiwan, between January 2007 and December 2010.

Exclusion Criteria:

* Cases in which estradiol levels exceeded 50 pg/mL on the second day of the menstrual cycle were excluded.
* Female minors or disabled persons.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with different causes of infertility
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate of intracytoplasmic sperm injection and laser assisted hatching on in vitro fertilization outcomes of patients with different causes of infertility | 3 months

SECONDARY OUTCOMES:
Live birth rate of intracytoplasmic sperm injection and laser assisted hatching on in vitro fertilization outcomes of patients with different causes of infertility | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan